CLINICAL TRIAL: NCT02698696
Title: Validation of a Cognitive Remediation Program for Bipolar Disorders
Acronym: ECO-BIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Clémence ISAAC, Psychologist, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 10477M
Record Dates: First submitted 2016-02-12; First posted 2016-03-04 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Bipolar Disorder
Keywords: Cognitive Remediation; Mood disorders; Neuropsychology
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ECo program (Experimental): Objective: to inform the patient about cognitive impairments and their repercussions; to train the patient in problem-solving skills through exercises; to implement strategies in daily life Duration: three months Frequency: two one-hour individual sessions and one hour of at-home training per week Modalities: pen and paper exercises, tools (tokens, cards, maps, chessboard) Modules: Psychoeducation, Attention, Memory, Executive Functions, Functional Impairments
  Interventions: Other: ECo program
- CRT program (Experimental): Objective: problem-solving skills training through exercises, in order to use strategies in daily life Duration: three months Frequency: two one-hour individual sessions and one hour of at-home training per week Modalities: pen and paper exercises Modules: Cognitive Flexibility, Working Memory, Planning
  Interventions: Other: CRT program
- Supportive psychotherapy (Active Comparator): Individual psychotherapy sessions focussing on autonomy in daily life, management of mood disorders' cognitive and functional impact, social skills, and the regulation of sleep and daily activities.
  Interventions: Other: Supportive psychotherapy

INTERVENTIONS:
Other: ECo program
  Arms: ECo program
Other: CRT program
  Arms: CRT program
Other: Supportive psychotherapy
  Arms: Supportive psychotherapy

SUMMARY:
This study evaluates the effect of a new cognitive remediation program designed for patients suffering from a bipolar disorder, on cognitive functions, psychosocial functioning and neural processes. In this double-blind (patient, outcomes assessor) controlled randomized trial the investigators compare patients receiving the ECo program for bipolar disorders, to patients benefiting from the broadly used cognitive remediation program CRT and to patients receiving supportive psychotherapy. Patients are treated for 3 months and monitored for 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Type I or type II Bipolar Disorder diagnosis, according to DSM-IV-TR criteria
2. No Manic or Major Depressive episode during the last three months
3. No or few residual depressive symptoms (HDRS-17 ≤ 12)
4. No or few residual manic symptoms (YMRS ≤ 8)
5. Stable dose of medication for the last two months
6. Cognitive complaint expressed by the patient and impairment observed by the patient's regular psychiatrist
7. Informed consent form read, initialed and signed
8. Patient registered on the social welfare system

Exclusion Criteria:

1. Other diagnosis than Bipolar Disorder on axis I of the DSM-IV-TR
2. Rapid Cycling Bipolar Disorder diagnosis
3. Addiction or substance abuse (except tobacco) during the twelve last months
4. Physical or neurological disorder that can lead to cognitive impairment
5. Engagement in a research protocol either currently or over the last month
6. Neuropsychological assessment or Rorschach Inkblot Test evaluation during the last six months
7. Ineligibility for Magnetic Resonance Imaging [MRI] (e.g. claustrophobia, metallic implants, pace-maker, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Perceptual Reasoning Index at 3 months | baseline and 3 months
  Composite score of the Wechsler Adult Intelligence Scale - fourth edition
Change from 3-months Perceptual Reasoning Index at 9 months | 3 months and 9 months
  Composite score of the Wechsler Adult Intelligence Scale - fourth edition

SECONDARY OUTCOMES:
Working Memory Index | baseline, 3 months and 9 months
  Composite score of the Wechsler Adult Intelligence Scale - fourth edition
Processing Speed Index | baseline, 3 months and 9 months
  Composite score of the Wechsler Adult Intelligence Scale - fourth edition
Rey Auditory Verbal Learning Test | baseline, 3 months and 9 months
  Neuropsychological test assessing verbal memory
Cardebat's Verbal Fluencies | baseline, 3 months and 9 months
  Neuropsychological test
Emotion Hexagon | baseline, 3 months and 9 months
  Task from the Facial Expressions of Emotion: Stimuli and Tests scale, assessing the recognition of emotions on faces
Key Search Test | baseline, 3 months and 9 months
  Task from the Behavioral Assessment of the Dysexecutive Syndrome scale, assessing planing abilities
Stroop Color Word Test | baseline, 3 months and 9 months
  Neuropsychological test assessing inhibition abilities
Hamilton Depression Rating Scale | 15 days before baseline, 3 months and 9 months
Young Mania Rating Scale | 15 days before baseline, 3 months and 9 months
Functional Repercussions Scale | baseline, 3 months and 9 months
  Self-assessment scale evaluating the consequences of cognitive impairments in daily life
Social Desirability Scale | baseline, 3 months and 9 months
  Self-assessment scale
Social Relationships Scale | baseline, 3 months and 9 months
  Self-assessment scale
Self-Appraisal of Illness Questionnaire | baseline, 3 months and 9 months
  Self-assessment scale
Rorschach Inkblot Test | baseline, 3 months and 9 months
Change from baseline Event-Related Potentials [ERP] P300 at 3 months during an Oddball task | baseline and 3 months
  Assessed for the first third of included patients
Change from baseline Event-Related Potentials [ERP] N2/P3 complex at 3 months during an emotional Stroop task | baseline and 3 months
  Assessed for the first third of included patients
Change from baseline serum Brain-Derived Neurotrophic Factor [BDNF] level (ng/mL) at 3 months | baseline and 3 months
  Assessed for the second third of included patients
Change from baseline functional Magnetic Resonance Imaging frontal activation at 3 months during an emotion recognition task | baseline and 3 months
  Assessed for the last third of included patients

CONTACTS AND LOCATIONS:
Overall Officials: Clémence Isaac, Psychologist, Principal Investigator — Unité de Recherche Clinique, EPS Ville Evrard
Locations (1):
- Unité de Recherche Clinique, EPS Ville Evrard, Neuilly-sur-Marne, France

REFERENCES:
- [Background] Altshuler LL, Ventura J, van Gorp WG, Green MF, Theberge DC, Mintz J. Neurocognitive function in clinically stable men with bipolar I disorder or schizophrenia and normal control subjects. Biol Psychiatry. 2004 Oct 15;56(8):560-9. doi: 10.1016/j.biopsych.2004.08.002. PMID 15476685
- [Result] Deckersbach T, Nierenberg AA, Kessler R, Lund HG, Ametrano RM, Sachs G, Rauch SL, Dougherty D. RESEARCH: Cognitive rehabilitation for bipolar disorder: An open trial for employed patients with residual depressive symptoms. CNS Neurosci Ther. 2010 Oct;16(5):298-307. doi: 10.1111/j.1755-5949.2009.00110.x. PMID 19895584
- [Result] Martinez-Aran A, Torrent C, Sole B, Bonnin CM, Rosa AR, Sanchez-Moreno J, Vieta E. Functional remediation for bipolar disorder. Clin Pract Epidemiol Ment Health. 2011;7:112-6. doi: 10.2174/1745017901107010112. Epub 2011 Jun 6. PMID 21687565